CLINICAL TRIAL: NCT02544490
Title: Defining Circulating Micro-RNA Biomarkers for the Early Diagnosis and Prognosis of Sepsis
Acronym: miRNA-Sepsis
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); MiRXES Pte Ltd (Industry); A*Star (Other)
Responsible Party: Principal Investigator, Emergency, Senior Consultant, National University Hospital, Singapore
Other Study IDs: TA/0029/2014
Record Dates: First submitted 2015-08-29; First posted 2015-09-09 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Sepsis
Keywords: Sepsis; MicroRNAs; Diagnosis; Prognosis
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood extraction from subjects subsequently separated to plasma and serum that are stored in the Tissue Repository.
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives are to:

1. derive and validate a panel of miRNAs that are consistently differentially expressed in the plasma of patients with and without sepsis
2. investigate the prognostic and predictive values of the panel of miRNAs to guide treatment
3. investigate the roles of these differentially-expressed circulating miRNAs in immune modulation during sepsis

The methodology involves sampling of blood from controls and subjects in the sepsis continuum at their earliest presentation in the emergency department longitudinally to hospitalization. The investigators will develop panels of miRNAs that are specific to early and late stages of sepsis, and correlate clinical, biochemical and microbiological outcomes with these miRNAs.

DETAILED DESCRIPTION:
Prospective observational cohort of patients along the entire sepsis continuum in National University Hospital Emergency Department (ED) will be enrolled along with non-infective controls. Whole blood samples will be separated immediately into plasma and serum for storage at the Tissue Repository. Those who are subsequently admitted to the general ward, high dependency (HD) or intensive care unit (ICU) will have their 2nd and 3rd samples obtained at 24-48 hours and 48-72 hours respectively. The 2nd and 3rd samples will be used as prognostic markers (Objective #2). Patients who are discharged directly from the ED will be tracked for any clinical recurrence of their disease within 28 days to ensure the diagnostic accuracy of the first sample of biomarkers that are extracted.

Samples will be batch-processed via the circulating miRNA profiling workflow comprising of the pre-analytics, analytics, and data processing and analysis phases. This qPCR-based miRNA profiling has much smaller feature to sample ratio thus allowing a global sequential forward selection to optimally combine a host of features with complementary prediction strengths to form the biomarker panel which has the least number of components and the maximized classification power (ROC AUC). Panel robustness measurement using computational generated noises and validation with a larger set of blinded samples will be performed.

The final objective will be assessed by measuring the concentrations of secreted cytokines, chemokines and reactive oxygen species after synthesis and transfection the newly-derived miRNA panel into monocytes and monocytic cell lines.

ELIGIBILITY:
Inclusion criteria for controls:

* Adults 21 years and above
* Has condition unrelated to any infective cause

Exclusion criteria for controls:

* Underlying chronic inflammatory condition (e.g. inflammatory bowel disease)
* Underlying autoimmune disease (e.g. rheumatoid arthritis, systemic lupus erythematosus)
* Pre-existent immunological disorder

Inclusion criteria for subjects:

* Adults 21 years and above
* Clinical/radiological suspicion or confirmation of infection

Exclusion criteria for subjects:

* Age below 21 years
* Prisoners
* Known pregnancy
* Do-not-attempt resuscitation status
* Requirement for immediate surgery
* Active chemotherapy
* Hematological malignancy
* Treating physician deems aggressive care unsuitable
* Unable to provide informed consent or comply with study requirements

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research project will be a prospective observational cohort study of controls without infection and patients along the entire sepsis continuum the Emergency Department (ED). Admitted patients will be followed-up in the inpatient units including the intensive care unit (ICU) and general wards. Healthy controls and those with systemic inflammatory response syndrome (SIRS) but without evidence of infection will also be recruited to demonstrate differentiation of biomarkers for early diagnosis. The reference standards for infection and sepsis will be positive cultures (e.g. from blood, urine, endotracheal tube, sputum) and final discharge diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Fold changes of miRNA expression | 3 years
  Fold changes of differentially-expressed miRNA in log2 scale in comparison to the severity of sepsis (control vs. sepsis vs. septic shock) and adjudicated requirement for hospitalization (yes vs. no)

SECONDARY OUTCOMES:
MiRNA panel test performance metrics | 3 years
  Sensitivity, specificity and likelihood ratios of capability of miRNA panel to distinguish different severity of sepsis (i.e. requirement for inpatient management) and against standard clinical parameters, C-reactive protein, procalcitonin, and inflammatory cytokines (interleukin-6, interleukin-8).

CONTACTS AND LOCATIONS:
Overall Officials: Win Sen Kuan, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore